CLINICAL TRIAL: NCT05949021
Title: OCTANE: Adjuvant Liposomal Doxorubicin and Carboplatin for Early-stage Triple Negative Breast Cancer
Brief Title: OCTANE: Adjuvant Liposomal Doxorubicin and Carboplatin for Early-stage Triple-negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mridula George, MD (Other)
Responsible Party: Sponsor-Investigator, Mridula George, MD, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 042304; Pro2023001280 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2023-07-06; First posted 2023-07-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Triple Negative Breast Cancer (TNBC)
Keywords: Liposomal doxorubicin; Carboplatin; Triple negative breast cancer (TNBC); Adjuvant therapy; Multicenter; Phase II clinical trial
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Liposomal doxorubicin and Carboplatin (Experimental): Combination of liposomal doxorubicin 30milligrams per square meter (mg/m2) and carboplatin area under the curve 5 (AUC 5), administered every four weeks for four cycles.
  Participants with triple-negative breast cancer (TNBC):
  1. Completed breast surgery and sentinel lymph node biopsy
  2. Tumor size less than2.5 and NO/ N1mi disease
  Interventions: Drug: Combination of liposomal doxorubicin

INTERVENTIONS:
Drug: Combination of liposomal doxorubicin — Combination of liposomal doxorubicin 30 milligrams per square meter and carboplatin (area under the curve 5), administered every 4 weeks for 4 cycles.

SUMMARY:
This clinical trial aims to evaluate the efficacy, safety, and exploratory measures of liposomal doxorubicin and carboplatin combination therapy in the adjuvant setting for early stage triple negative breast cancer (TNBC) patients.

The primary objective is to determine the effectiveness of liposomal doxorubicin and carboplatin in reducing the risk of recurrence for early stage TNBC patients.

The secondary objectives involve characterizing the safety and toxicity profile of the combination therapy. Adverse events rates will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

The exploratory objectives of the study focus on evaluating changes in circulating tumor DNA (ctDNA). This measure will provide insights into the potential utility of ctDNA as a biomarker for treatment response and disease progression.

By addressing these objectives, the study aims to contribute to the understanding of the benefits and risks associated with liposomal doxorubicin and carboplatin combination therapy in the adjuvant setting for early stage TNBC, potentially leading to improved treatment outcomes and patient care.

DETAILED DESCRIPTION:
Background Triple negative breast cancer (TNBC) is a subtype of breast cancer characterized by the absence of estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor 2 (HER2) expression. TNBC is associated with a higher risk of recurrence and poorer prognosis compared to other breast cancer subtypes. Currently, the standard of care for early stage TNBC includes adjuvant chemotherapy, typically consisting of anthracyclines and taxanes. However, this regimen is associated with significant toxicities and adverse effects.

This clinical trial aims to evaluate the combination of liposomal doxorubicin and carboplatin as an adjuvant therapy for patients with early stage TNBC. Previous studies conducted in the neoadjuvant setting have shown promising results with this combination, indicating a reduction in the risk of recurrence. Additionally, the combination has demonstrated a more favorable tolerability profile compared to the current standard of care. Therefore, this trial seeks to assess the efficacy and safety of liposomal doxorubicin and carboplatin in the adjuvant setting for TNBC.

The primary objective of this clinical trial is to determine the efficacy of liposomal doxorubicin and carboplatin as adjuvant therapy for early stage TNBC. The efficacy will be measured by evaluating the recurrence-free survival (RFS) rate at a specified time point.

The secondary objectives of this study include: Characterizing the safety and toxicity profile of the combination therapy, as measured by the incidence and severity of adverse events using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Assessing the overall survival (OS) rate in patients receiving liposomal doxorubicin and carboplatin. Evaluating the pathological complete response (pCR) rate following the treatment regimen. Analyzing the disease-free survival (DFS) rate in patients treated with the combination therapy. In addition to the primary and secondary objectives, this study also aims to explore the following: Investigating changes in circulating tumor DNA (ctDNA) levels as a potential biomarker for treatment response and disease progression. Exploring correlations between specific genetic markers and treatment outcomes.

This study is a multicenter, open-label, phase II clinical trial. The study will enroll patients with early stage TNBC who have undergone surgical resection of the primary tumor. Patients in the study will receive adjuvant therapy consisting of liposomal doxorubicin and carboplatin. The dosing and administration schedule will be determined based on established guidelines and previous studies.

The sample size calculation will be based on statistical considerations, taking into account the primary endpoint of recurrence-free survival. A predetermined number of patients will be required to achieve adequate statistical power.

Eligible patients will be enrolled and undergo baseline assessments, including medical history, physical examination, laboratory tests, and imaging studies. Treatment will be initiated according to the predetermined dosing and administration schedule. Patients will be closely monitored throughout the study for treatment response, adverse events, and disease recurrence.

Follow-up visits will be scheduled at specified time intervals to assess long-term outcomes and collect additional data.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed early stage triple negative breast cancer (TNBC) with a primary tumor size less than 2.5cm and nodal disease of N0/N1mi on final surgical pathology.
* Patients who have completed primary surgical treatment.
* Estrogen receptor (ER) expression of 20% or less, progesterone receptor (PgR) expression of 20% or less, and human epidermal growth factor receptor 2 (HER2) status 0-2+ by immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH) result of 2.0 or less.
* Participants with a history of prior cancers are allowed if there is no evidence of disease within the last five years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Baseline left ventricular ejection fraction (LVEF) greater than 50% (most recent measurement within the last 5 years).
* No prior history of treatment with anthracycline-based chemotherapy.
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) greater than or equal to 1500/uL.
  * Platelet count greater than or equal to 100,000/uL.
  * Hemoglobin level greater than or equal to 9.0 g/dL.
* Adequate hepatic function:

  * Total bilirubin less than or equal to 1.5 times the upper limit of normal (ULN).
  * Aspartate aminotransferase (AST) levels (also known as serum glutamic-oxaloacetic transaminase, SGOT) less than or equal to 5 times the ULN.
  * Alanine aminotransferase (ALT) levels (also known as serum glutamic-pyruvic transaminase, SGPT) less than or equal to five times the ULN.
  * Participants with biliary obstruction must have restored biliary flow through the placement of an endoscopic common bile duct stent or percutaneous drainage.
* Adequate renal function, with a creatinine level less than 1.5 times the institutional ULN or a calculated creatinine clearance greater than or equal to 50 mL/min using the Cockcroft-Gault formula.
* Ability to understand the nature of the study protocol and provide written informed consent.
* Willingness and ability to comply with scheduled visits and treatment plans.

Exclusion Criteria:

* Participants with stage III-IV breast cancer.
* Uncontrolled hypertension, defined as systolic blood pressure greater than 190 mm Hg or diastolic blood pressure greater than 100 mm Hg.
* Active liver disease.
* Any condition, including the presence of laboratory abnormalities that, in the investigator's opinion, would place the participant at an unacceptable risk if they were to participate in the study.
* Pre-existing sensory neuropathy greater than grade 1.
* Clinically significant cardiac disease, such as congestive heart failure, symptomatic coronary artery disease, and uncontrolled cardiac arrhythmias, or a history of myocardial infarction within the last six months.
* Presence of a serious non-healing wound, ulcer, or bone fracture.
* Participants with uncontrolled and/or active infection with HIV, Hepatitis B, or Hepatitis C.
* Participants with a history of allergy or hypersensitivity to any of the study drugs.
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women
Enrollment: 30 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) Rate | From the start of the study up to 5 years
  The disease-free survival (DFS) rate is used to evaluate the efficacy of liposomal doxorubicin and carboplatin in the adjuvant setting. It assesses the proportion of participants who remain free from disease recurrence or progression after receiving the combination treatment as an adjuvant therapy for their cancer.
  DFS rate is calculated by dividing the number of participants who have not experienced disease recurrence or progression within a specified timeframe by the total number of participants enrolled in the clinical trial.
  DFS Rate (%) = (Number of participants with no disease recurrence or progression / Total number of participants enrolled) × 100 A higher DFS rate indicates a greater efficacy of liposomal doxorubicin and carboplatin as an adjuvant treatment, suggesting their ability to delay or prevent disease recurrence or progression in participants. A higher DFS rate implies a better prognosis and improved disease control in the adjuvant setting.

SECONDARY OUTCOMES:
Safety and Toxicity Profile of the Study Treatment as measured by Adverse Events Rates and Common Terminology Criteria for Adverse Events version 5 (CTCAE v.5) | From the start of the study up to 5 years
  The outcome measure aims to characterize the safety and toxicity profile of the study treatment by assessing the occurrence and severity of adverse events (AEs) as measured using the CTCAE v.5). The CTCAE v.5 utilizes a standardized grading scale to assess the severity of adverse events. The scale consists of grades ranging from 1 to 5, with each grade corresponding to a specific level of severity. The grades are:
  Grade 1 Mild Event is asymptomatic or mild, requiring minimal or no medical intervention.
  Grade 2 Moderate Event minimal to moderate interference with daily activities, and some medical intervention.
  Grade 3 Severe Event causes significant interference with daily activities, and medical intervention or treatment is required.
  Grade 4 Life-threatening or disabling Event poses immediate risk to life or function, requiring urgent medical intervention or treatment.
  Grade 5 Death Event results in death related to the adverse event.

OTHER OUTCOMES:
Changes in Circulating Tumor DNA (ctDNA) Levels. Monitoring ctDNA Dynamics Pre and Post Treatment | Baseline and (on cycle four) at sixteen weeks,6,12,18,24 months up to five years post treatment
  The outcome measure aims to evaluate changes in circulating tumor DNA (ctDNA) levels as a marker of treatment response. It involves monitoring and comparing the levels of ctDNA before and after the administration of the treatment to assess the impact of the treatment on tumor burden and disease progression.
  The levels of ctDNA will be measured at multiple time points, including baseline (pre-treatment) and post-treatment intervals. This can be done using various techniques such as next-generation sequencing (NGS) or polymerase chain reaction (PCR) assays targeting specific tumor-associated genetic alterations. The quantitative analysis of ctDNA will provide insights into the changes in tumor burden and the potential efficacy of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mridula George, MD, Principal Investigator — Cancer Institute of New Jersey Rutgers
Locations (8):
- United States (8):
  - RWJBarnabas Health - Trinitas hospital and Comprehensive Center, Elizabeth, New Jersey
  - RWJBarnabas Health Jersey City Medical Center, Jersey City, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - RWJBarnabas Health - Newark Beth Israel Medical Center, Newark, New Jersey
  - University Hospital-Newark, Newark, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No